CLINICAL TRIAL: NCT02560506
Title: Development of Low Cost Devices to Increase Access to Treadmill Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, T. George Hornby, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Model Systems
Record Dates: First submitted 2015-09-15; First posted 2015-09-25 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elastic assisted treadmill walking (Experimental): Participants will participate in treadmill training with a low cost pulley system device made of rubber bands (Theraband(R)), which will assist therapists in advancing limbs while gait training.
  Interventions: Device: Elastic assisted treadmill walking

INTERVENTIONS:
Device: Elastic assisted treadmill walking — Rubber band pulley system that will assist therapists in advancing limbs while gait training. The device is positioned in front of a treadmill and the stretch of the elastic bands when a legs moves backwards on a treadmill is resists the movement and facilitates limb swing when walking.
  Other Names: Theraband(R)

SUMMARY:
The goals of this Model System Program are to expand upon and advance the findings and outcomes of previous and current Model Systems clinical research, to continue to develop and study the effectiveness of innovative treatment strategies for persons with spinal cord injury (SCI); and to evaluate the benefits of a well-designed, comprehensive, coordinated, interdisciplinary continuum of care that lead to improved outcomes for all persons with SCI. In order to achieve these goals, the following objectives of the Midwest Regional Spinal Cord Injury Care System (MRSCICS) model system grant proposal will be accomplished.

DETAILED DESCRIPTION:
The investigators will develop and assess the use of spring-loaded devices to assist limb swing and forward propulsion during body weight supported treadmill training (BWSTT) (Aim 1). Prototype models of both devices have been developed.

These devices will be:

1. simple to use in the clinical setting;
2. will be easily adjustable to alter the assistance provided; and,
3. will be able to quantify the amount of assistance necessary to facilitate normal stepping patterns.

The investigators will also evaluate short- and long-term adaptations in locomotor performance following BWSTT in individuals with incomplete SCI with the use of these devices. This information will identify the effects of variable assistance at the limbs or trunk to modulate muscle activity and/or motor performance (kinematics) during stepping to maximize walking recovery.

ELIGIBILITY:
Inclusion Criteria:

* non-progressive lesion between spinal levels C1-T10 of > 3 months duration. Subjects with below T10 will be excluded due to potential lower motor neuron (LMN) injury
* score > 10 on the Lower Extremity Motor Score (LEMS) developed previously to measure strength in SCI. For the LEMS criteria, preliminary data indicate that subjects with LEMS < 10 in the chronic stages do not recover walking
* All subjects must require physical assistance to ambulate on the treadmill at a speed of 4.0 kmph at 0% body weight support (BWS)
* All subjects will have an overground gait speed <.8m/s
* range of motion (ankle: -10 to 30 deg, knee: 0 to 90 deg, hip: -10 to 40 deg) consistent with gait
* medically stable with medical clearance to participate (absence of concurrent illness, including unhealed decubiti, infection, cardiopulmonary disease, osteoporosis, active heterotrophic ossification or peripheral nerve damage in the lower limbs, history of traumatic head injury)
* able to tolerate 30 minutes of upright (standing) position without orthostasis (decrease in blood pressure by 20 mmHg systolic and 10 mmHg diastolic; minimized with ambulatory population)
* women of childbearing potential

Exclusion Criteria:

* women who are pregnant will be excluded due to potential forces at trunk from BWS or pelvic assistance
* those in concurrent physical therapy to eliminate effects of additional interventions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in locomotor performance during treadmill walking | outcomes will be assessed prior to and following up to 8 weeks of training
  Evaluation of the changes in treadmill speed (m/s) prior to and following use of the device

SECONDARY OUTCOMES:
Change in oxygen consumption | outcomes will be assessed prior to and following up to 8 weeks of training
  Metabolic costs (oxygen ml/kg/min) will be collected using a portable metabolic system (K4b2 , CosMed USA, Inc., Chicago) during treadmill training in both groups

OTHER OUTCOMES:
Changes in overground gait speed | outcomes will be assessed prior to and following up to 8 weeks of training
  Gait speed (m/s) will be collected during overground walking

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Hornby, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States